CLINICAL TRIAL: NCT05029726
Title: Randomized, Placebo-controlled Trial of Erector Spinae Plane Blocks (ESPB) for Perioperative Pain Management for Minimally Invasive (MIS) Lumbar Spine Surgery
Brief Title: Regional Anesthesia in Minimally Invasive Lumbar Spine Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: John O'Toole (Other)
Responsible Party: Sponsor-Investigator, John O'Toole, Professor of Neurosurgery, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORA20050502
Record Dates: First submitted 2021-08-14; First posted 2021-08-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Disc Herniation; Lumbar Spondylolisthesis; Lumbar Spondylosis; Lumbar Radiculopathy; Lumbar Spine Instability; Synovial Cyst; Degenerative Disc Disease; Degenerative Spondylolisthesis; Degenerative Intervertebral Discs
Keywords: erector spinae plane block; minimally invasive spine surgery; regional anesthesia; randomized controlled trial
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Displacement; Spondylolisthesis; Spondylosis; Radiculopathy; Synovial Cyst; Intervertebral Disc Degeneration | interventions — Clonidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: All patients will undergo surgery using an enhanced recovery after surgery (ERAS) multi-modal anesthesia protocol that is currently in standard use for MIS lumbar spine surgical procedures. Patients will be randomized in a 1:1 ratio to investigational and control arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, surgeons and anesthesiologists will all be blinded to treatment allocation. Syringes containing the fluid to be injected will be prepared by pharmacy and labeled with subject number in such a manner to blind the anesthesiologist performing the ESPB to its contents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Investigational (Experimental): Patients will undergo regional ESPB with bupivacaine plus clonidine in the holding area of the OR immediately prior to surgery. 30mL of 0.25% bupivacaine/1:200,000 epinephrine/50mcg clonidine will be administered bilaterally (total 60ml) to the lumbar paraspinal erector spine plane using ultrasound-guidance.
  Interventions: Drug: Bupivacaine-Epinephrine 0.25%-1:200,000 Injectable Solution plus clonidine
- Control (Placebo Comparator): Patients will receive a placebo injection of normal saline via the same ESPB technique. 30ml of normal saline will be administered bilaterally (total 60ml) to the lumbar paraspinal erector spine plane using ultrasound-guidance.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Bupivacaine-Epinephrine 0.25%-1:200,000 Injectable Solution plus clonidine — Bupivacaine-Epinephrine 0.25%-1:200,000 plus clonidine 50 micrograms in 30cc syringes administered as ESPB
  Arms: Investigational
Drug: normal saline — normal saline in 30cc syringes administered using ESPB technique
  Arms: Control

SUMMARY:
Opioid overuse is a widespread public health crisis in the United States with increasing rates of addiction and overdose deaths from prescription opioids. Reducing the need for opiate analgesics in the post-operative setting has become a high priority in minimizing long-term opioid use in surgical patients. This study will serve to demonstrate the efficacy of the addition of regional analgesic techniques in reducing post-operative opioid requirements in patients undergoing common lumbar spinal surgical procedures.

DETAILED DESCRIPTION:
Opioid abuse and misuse remain a public health crisis in the United States, notably in patients with chronic pain from degenerative spine disease. Perioperative pain management for patients undergoing spinal surgery remains largely reliant on opioid medications, with several known adverse effects including, but not limited to delirium, postoperative urinary retention (POUR), constipation and nausea. These side effects contribute to increased hospital length of stay (LOS) with increased incidence of overall in-hospital complications, perioperative costs, and increased rates of opioid habituation and addiction.

Dependence on prescription opioids has been associated with wide-ranging social and economic consequences including increased opioid overdose resulting in death, growing opioid-related incarcerations, and spiraling opioid-related healthcare cost from treatment of addiction, opioid-related mental health issues, and debilitating chronic pain. Long-term requirements for opioid medications may be associated with the use of higher doses of opioids in the perioperative period for patients undergoing invasive surgery for spinal degenerative conditions. Studies have demonstrated that patients who consume fewer opioids for 30 days after surgery are less likely to progress to become chronic opioid users. Regional analgesic techniques have shown promise in decreasing post-operative pain and opioid requirements in thoracic and abdominal surgery but difficulties with post-operative neurological assessments have limited their use in spinal surgery. Inter-fascial plane blocks, however, have emerged as a safe and potentially useful regional analgesic technique to mitigate the pain-inducing effects of posterior spine surgery.

Erector Spinae Plane Blocks (ESPBs), specifically, involve ultra-sound guided injection of local anesthetic (LA) posteriorly beneath the erector spinae muscles resulting in longitudinal and ventrolateral spread of the anesthetic into the paravertebral space where the ventral and dorsal rami of the spinal nerves are located thereby inducing a multi-level analgesic effect. Depending upon the LA used, this effect may last for 4 to 36 hours.

The proposed study will examine the efficacy of preoperative ESPBs in reducing post-operative opioid utilization and its associated complications specifically after minimally invasive (MIS) lumbar spine surgery including both decompressive and instrumented fusion procedures. The guiding principle of MIS spine surgery is reduction of iatrogenic injury by utilizing muscle dilating approaches and tubular retractors rather than conventional open, subperiosteal muscle stripping techniques. The latter typically results in muscle denervation and devascularization as well as postoperative muscle atrophy and dead space creation that increase postoperative pain, muscle dysfunction, prolonged recovery times and complications. Since MIS spinal surgical procedures preserve normal paraspinal musculature compared to open surgery, the magnitude of effect of ESPBs may actually be more pronounced in this population.

The investigators hypothesize that by conducting this investigation within the rigor of a double-blinded, randomized placebo-controlled clinical trial, the results will definitively demonstrate that the addition of regional analgesia in the form of ESPB during MIS lumbar spine surgery will 1) reduce post-operative opioid consumption and 2) reduce opioid-related complications and hospital LOS but 3) have no adverse effects on postoperative pain control.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Undergoing one of 3 procedure types: 1) 2 or more levels of MIS decompression (e.g., discectomy, foraminotomy, laminectomy); 2) 1-3 levels of MIS transforaminal lumbar interbody fusion (TLIF) (with or without additional levels of MIS decompression for no greater than 3 total operative levels); 3) 1-3 levels of anterior lumbar interbody fusion (ALIF) or MIS lateral lumbar interbody fusion (LLIF) accompanied by posterior percutaneous instrumentation at the same levels
* Willing and able to give consent

Exclusion Criteria:

* Opioid tolerant at the time of the surgical procedure--defined as consuming greater than 30mg of morphine milligram equivalents (MME) daily (https://www.cdc.gov/drugoverdose/prescribing/guideline.html)
* Presence of an indwelling pain device (e.g., intrathecal opioid pump, spinal cord stimulator, dorsal root ganglion stimulator)
* Known allergy to bupivacaine, clonidine or similar local anesthetics
* Indication for surgery other than degenerative disease (e.g., neoplasm, infection, trauma)
* Chronic kidney disease (stage 3 or greater), or hepatic failure
* Active pregnancy
* Disease process or mental illness that would preclude accurate evaluation of pain in the perioperative period
* Active Worker's Compensation litigation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Inpatient opioid consumption | Every 1 day during inpatient admission up to 30 days
  Mean per day inpatient opioid consumption in morphine milligram equivalents (MME)

SECONDARY OUTCOMES:
Post-discharge opioid consumption | 14 days (+/- 7days) ,56 days (+/- 14 days) and 90 days (+/- 19) postoperatively
  Total and per day mean postoperative opioid consumption after hospital discharge in MME as recorded in medication diary by patients
Postoperative opioid prescriptions filled | From hospital discharge to 90 days postoperatively
  • Total MMEs of opioid prescriptions filled as found on the Illinois Prescription Monitoring Program website
Length of hospital stay | From time of surgery to time discharge criteria met in hours, up to 2160 hours
  Duration of hospital stay postoperatively measured in days as determined by the time at which each patient met discharge criteria
Postoperative Urinary Retention (POUR) | Immediately post-surgery to discharge, up to 90 days
  Incidence of POUR measured as proportion of inpatient hospital days demonstrating the need for straight catheterization or foley placement
Post-operative delirium | Immediately post-surgery to discharge
  Incidence of post-operative delirium as measured by the need for placement of physical restraints
Post-operative delirium | Immediately post-surgery to discharge, up to 90 days
  Incidence of post-operative delirium as measured by the administration of new anti-psychotic medications
Postoperative pain scores | Every 1 day during inpatient admission up to 30 days
  Mean daily VAS (visual analog scale) pain scores recorded in the electronic medical record (EMR)
Patient-reported pain and functional outcomes | From baseline preoperative values to 6 week post-operative values
  Change in Visual Analog Scale (VAS) for pain in the back and leg (0-10 with 10 being worst)
Patient-reported pain and functional outcomes | From baseline preoperative values to 6 week post-operative values
  Change in Oswestry Disability Index (ODI; 0 to 100 with 100 being worst)
Patient-reported pain and functional outcomes | From baseline preoperative values to 6 week post-operative values
  Change in Short Form 12/6D (SF-12/6D; 0 to 100 with 0 being worst)
Peri-operative complications | Time of surgery to 6 weeks postoperative
  Prospectively documented medical and surgical complications/adverse events (AEs) including rates of readmission or reoperation for AEs

CONTACTS AND LOCATIONS:
Overall Officials: John O'Toole, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin KJ, Lewis S. Opioid-free Analgesia for Posterior Spinal Fusion Surgery Using Erector Spinae Plane (ESP) Blocks in a Multimodal Anesthetic Regimen. Spine (Phila Pa 1976). 2019 Mar 15;44(6):E379-E383. doi: 10.1097/BRS.0000000000002855. PMID 30180150
- [Background] Chin KJ, Dinsmore MJ, Lewis S, Chan V. Opioid-sparing multimodal analgesia with bilateral bi-level erector spinae plane blocks in scoliosis surgery: a case report of two patients. Eur Spine J. 2020 Dec;29(Suppl 2):138-144. doi: 10.1007/s00586-019-06133-8. Epub 2019 Sep 3. PMID 31482311
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Melvin JP, Schrot RJ, Chu GM, Chin KJ. Low thoracic erector spinae plane block for perioperative analgesia in lumbosacral spine surgery: a case series. Can J Anaesth. 2018 Sep;65(9):1057-1065. doi: 10.1007/s12630-018-1145-8. Epub 2018 Apr 27. PMID 29704223
- [Background] Singh S, Choudhary NK, Lalin D, Verma VK. Bilateral Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: A Randomized Control Trial. J Neurosurg Anesthesiol. 2020 Oct;32(4):330-334. doi: 10.1097/ANA.0000000000000603. PMID 31033625
- [Background] Ueshima H, Inagaki M, Toyone T, Otake H. Efficacy of the Erector Spinae Plane Block for Lumbar Spinal Surgery: A Retrospective Study. Asian Spine J. 2019 Apr;13(2):254-257. doi: 10.31616/asj.2018.0114. Epub 2018 Nov 15. PMID 30424594
- [Background] van den Broek RJC, van de Geer R, Schepel NC, Liu WY, Bouwman RA, Versyck B. Evaluation of adding the Erector spinae plane block to standard anesthetic care in patients undergoing posterior lumbar interbody fusion surgery. Sci Rep. 2021 Apr 7;11(1):7631. doi: 10.1038/s41598-021-87374-w. PMID 33828209
- [Background] Armaghani SJ, Lee DS, Bible JE, Archer KR, Shau DN, Kay H, Zhang C, McGirt MJ, Devin CJ. Preoperative opioid use and its association with perioperative opioid demand and postoperative opioid independence in patients undergoing spine surgery. Spine (Phila Pa 1976). 2014 Dec 1;39(25):E1524-30. doi: 10.1097/BRS.0000000000000622. PMID 25417827
- [Background] Kalakoti P, Hendrickson NR, Bedard NA, Pugely AJ. Opioid Utilization Following Lumbar Arthrodesis: Trends and Factors Associated With Long-term Use. Spine (Phila Pa 1976). 2018 Sep 1;43(17):1208-1216. doi: 10.1097/BRS.0000000000002734. PMID 30045343